CLINICAL TRIAL: NCT06368622
Title: A Post-Market Clinical Follow-up Study to Evaluate the Long-Term Safety and Effectiveness of Surpass Evolve Flow Diverter System
Brief Title: Evolve China PMCF Study
Status: Recruiting | Type: Observational
Sponsor: Stryker Neurovascular (Industry)
Collaborators: Stryker (Beijing) Healthcare Products Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CDM10001814
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Intracranial Aneurysm
Keywords: intracranial aneurysms; flow diverter system; Surpass Evolve Flow Diverter System; Surpass Evolve
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Surpass Evolve Flow Diverter System — Endovascular treatment with Surpass Evolve Flow Diverter System was performed in patients diagnosed with intracranial aneurysms

SUMMARY:
A prospective, multi-center, single-arm, open-label, observational, post-market clinical follow-up. The expected duration of the study is 8 years (including up to 5-years' follow-up). Each subject will be followed up per standard of care (SoC) at each study site.

ELIGIBILITY:
Inclusion Criteria:

* Subject age is ≥ 18 and ≤80 years
* Subject is eligible for Surpass Evolve FDS IFU, and/or physician intends to treat the subject with Surpass Evolve FDS per his/her judgement
* Subject, or subject's legally authorised representative (LAR) has provided signed informed consent using the Ethics Committee (EC)-approved consent form
* Subject is willing to comply with scheduled visits and examinations per institutional SOC

Exclusion Criteria:

* Subject has any non-target intracranial aneurysm treated within 30 days prior to study enrollment
* Subject has a planned treatment of a non-target aneurysm in the same vascular territory during participation in the study within 12 months post procedure
* Subject has undergone previous treatment where it would interfere with the delivery and/ or placement and/or proper apposition of Surpass Evolve FDS
* Subject has acute target aneurysm rupture and/or subarachnoid hemorrhage occurred within 30 days prior to enrollment
* Subject has any condition demonstrated as Warning or Precautions in IFU
* Antiplatelet and/or anticoagulation therapy (e.g. aspirin and clopidogrel) is contraindicated for the subject
* Subject has not received dual anti-platelet agents prior to the procedure
* Subject with an active bacterial infection
* Subject in whom the angiography demonstrates the anatomy is not appropriate for endovascular treatment, due to conditions such as:

  * Severe intracranial vessel tortuosity or stenosis; and/or
  * Intracranial vasospasm not responsive to medical therapy
* Female subjects who are pregnant/ nursing, or who are unwilling or unable to take adequate method of contraception prior to the 12-month study follow-up.*

  *If the subject becomes pregnant during her participation, the physician will have to evaluate the risk associated to her continuing participation to the rest of the study.
* Enrollment in another trial involving an investigational product and/or drug interfere with study procedure/ results
* The investigator determined that the health of the patient may be compromised by the patient's enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be enrolled from up to 40 study sites in China.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Neurological death or disabling stroke | 12 months (-3/ +6 months) post-procedure
  Neurological death or disabling stroke at 12 months post-procedure (-3/ + 6 months).
  * Neurological death defined as stroke-related death
  * Disabling stroke defined as stroke in the treated vascular territory that results in a mRS score ≥ 3, assessed by a qualified investigator at a minimum 90-days post stroke event
100% occlusion without significant parent artery stenosis | 12 months (-3/+6 months) post-procedure
  A composite of 100% occlusion (defined as Raymond-Roy class 1) of the target aneurysm without significant parent artery stenosis (significant stenosis defined as ˃50% stenosis), per the assessment of images required, and with no retreatment of target aneurysm at 12 months (-3/+6 months) post-procedure.

SECONDARY OUTCOMES:
Procedure- and device-related serious adverse events | 60 months
  Procedure- and device-related serious adverse events through 60 months post-procedure
Key neurological events | 60 months
  Key neurological events of interest through 60 months post-procedure
Procedural success | Intraprocedural
  Delivery and deployment of one or more study devices to completely cover the neck of the target aneurysm in an individual subject.
Device success | Intraprocedural
  Delivery and deployment of a study device to completely cover the neck of the target aneurysm, either alone or in conjunction with another Surpass Evolve FDS.
Re-sheathing success | Intraprocedural
  Successful re-sheathing with single attempt.

CONTACTS AND LOCATIONS:
Locations (22):
- China (22):
  - Xuanwu Hospital Capital Medical University, Beijing
  - Beijing Tiantan Hospital, Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing
  - Bethune First Hospital of Jilin University, Changchun
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Guangdong Second Provincial General Hospital, Guangzhou
  - First Affiliated Hospital of Kunming Medical University, Kunming
  - Nanyang Central Hospital, Nanyang
  - Ningbo Medical Center Lihuili Hospital, Ningbo
  - The Affiliated Hospital of Qingdao University, Qingdao
  - Shanghai Fourth People's Hospital Affiliated To Tongji University, Shanghai
  - South China Hospital of Shenzhen University, Shenzhen
  - The Eighth Affiliated Hospital, Sun Yat-sen University (Shenzhen Futian), Shenzhen
  - The Third Hospital of Hebei Medical University, Shijiazhuang
  - Tangshan Workers' Hospital, Tangshan
  - Tianjin Huanhu Hospital, Tianjin
  - Weifang People's Hospital, Weifang
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Xiangyang No.1 People's Hospital, Xiangyang
  - Zhuhai People's Hospital, Zhuhai
  - The Fifth Affiliated Hospital, Sun Yat-sen University, Zhuhai

IPD SHARING:
Plan to Share IPD: No